CLINICAL TRIAL: NCT04096014
Title: Late Evening and Early Morning Protein Supplement to Reduce Readmissions for Hepatic Encephalopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Srinivasan Dasarathy, Staff Physician, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18-749
Record Dates: First submitted 2019-09-11; First posted 2019-09-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Hepatic Encephalopathy
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ensure Enlive (Active Comparator)
  Interventions: Dietary Supplement: Ensure Enlive; Other: Standard Of Care
- Standard of Care (Placebo Comparator)
  Interventions: Other: Standard Of Care

INTERVENTIONS:
Dietary Supplement: Ensure Enlive — The subjects in the intervention group will receive two Ensure Enlive supplements per day for 180 days.
  Arms: Ensure Enlive
Other: Standard Of Care — The subjects in the Standard of care group will continue to receive the standard clinical therapy.

SUMMARY:
Readmission rates for patients with hepatic encephalopathy due to end stage liver disease are high. Hyperammonemia contributes significantly to encephalopathy and occurs because of impaired hepatic ureagenesis and increased skeletal muscle proteolysis. We propose a randomized, 6-month nutritional intervention in cirrhotic patients who have had at least 1 admission for hepatic encephalopathy within the last 6 months. We hypothesize that a combination of late evening and early morning protein supplement (Ensure Enlive) will decrease recurrent hepatic encephalopathy and consequent readmission rates by lowering skeletal muscle proteolysis and improved lean body mass.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* cirrhosis diagnosed by clinical history and liver biopsy and/or clinical, biochemical and imaging evidence of cirrhosis
* at least 1 hospitalization for documented HE within the last 12 months.
* abdominal CT scan anytime in the past

Exclusion Criteria:

* Patients with MELD score > 35
* end stage organ failure (major dysfunction requiring organ support)
* kidney injury defined by a creatinine > 2 mg/dl or rise in creatinine by 0.5 gm/dl from baseline that is unresponsive to withholding diuretics and intravenous albumin administration (1 gm/kg up to 100 gm/day)
* active malignancy
* uncontrolled diabetes mellitus with A1c>9.5 (to avoid altered muscle protein metabolism
* medications (anabolic steroids, corticosteroids) that affect skeletal muscle mass
* recent gastrointestinal surgery within past 12 months
* ongoing infection (positive blood or other body fluid cultures)
* active gastrointestinal bleeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Determine if decreasing nocturnal fasting by protein supplements will change readmission rates. | Day 0 & Day 180
  Change in number of readmissions

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No